CLINICAL TRIAL: NCT07102316
Title: A Phase 1, Open-Label, Randomized, 3-Group, Crossover Study to Assess the Relative Bioavailability After a Single Inhalation Administration of TPIP Formulation 2 (F2) to TPIP Formulation 3 (F3) in Healthy Participants
Brief Title: A Study to Assess the Relative Bioavailability After a Single Inhalation Administration of Treprostinil Palmitil Inhalation Powder (TPIP) Formulation 2 (F2) to TPIP Formulation 3 (F3) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INS1009-103
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TPIP Dose A (Experimental): Participants will receive single dose of TPIP F2 or F3 on Day 1 in treatment period 1 followed by single dose of TPIP F3 or F2 on Day 1 in treatment period 2. Both treatment periods are separated by 7-day washout period.
  Interventions: Drug: TPIP F2; Drug: TPIP F3
- TPIP Dose B (Experimental): Participants will receive single dose of TPIP F2 or F3 on Day 1 in treatment period 1 followed by single dose of TPIP F3 or F2 on Day 1 in treatment period 2. Both treatment periods are separated by 7-day washout period.
  Interventions: Drug: TPIP F2; Drug: TPIP F3
- TPIP Dose C (Experimental): Participants will receive single dose of TPIP F2 or F3 on Day 1 in treatment period 1 followed by single dose of TPIP F3 or F2 on Day 1 in treatment period 2. Both treatment periods are separated by 7-day washout period.
  Interventions: Drug: TPIP F2; Drug: TPIP F3

INTERVENTIONS:
Drug: TPIP F2 — Inhalation using a capsule-based dry powder inhaler device.
  Other Names: INS1009
Drug: TPIP F3 — Inhalation using a capsule-based dry powder inhaler device.
  Other Names: INS1009

SUMMARY:
The primary objective of this study is to determine the relative bioavailability of treprostinil (TRE) between the TPIP F2 and TPIP F3 at 3 capsule strengths, dose A, dose B, and dose C, in healthy participants following a single inhalation of TPIP dose.

ELIGIBILITY:
Inclusion Criteria

* Body mass index (BMI): 18.0 to 32.0 kilogram per square metre (kg/m^2), inclusive, at screening.
* Weight: ≥50 kg (kilograms), inclusive, at screening.
* Must be a nonsmoker (no use of tobacco or nicotine products) and/or has not used chewing tobacco for at least 1 month prior to screening.
* Participants must be able to inhale study treatment using a dry powder inhaler.
* All medication (including over-the-counter medication, health supplements such as St. John's wort extract) must have been stopped at least 14 days prior to clinical site admission. An exception is made for acetaminophen, which is allowed up to admission to the clinical facility. Female participants may continue to use hormonal contraceptives throughout the study.

Exclusion Criteria

* Female participants who are pregnant, nursing, or planning to become pregnant during the study.
* Participant has a positive serology test result for human immunodeficiency virus 1 or 2, hepatitis C virus antibodies, or hepatitis B surface antigen or hepatitis B core antibodies at screening. A positive result for hepatitis C virus antibodies will be allowed, if the participant has documented proof of prior, successful treatment.
* History of malignancy within 5 years prior to screening, with exception of completely treated in situ carcinoma of the cervix, and completely treated non-metastatic squamous cell or basal cell carcinoma of the skin.
* Use of drugs that inhibit or induce Cytochrome P2C8 (CYP2C8) within 3 weeks prior to first dose until follow-up visit.
* Participant has received any study drug in another investigational study within 30 days of screening or less than 5 times the drug's half-life, whichever is longer.
* QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 milliseconds (ms).
* The participant had active liver disease or hepatic dysfunction at screening or admission, manifested as:

  * Elevated liver function test results (Alanine Aminotransferase [ALT] or Aspartate Aminotransferase [AST] > 2 × Upper Limit of Normal [ULN])
  * Bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN; ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%)
  * Known hepatic or biliary abnormalities (excluding Gilbert's syndrome or asymptomatic gallstones)
* Participant has a platelet count less than lower limit of normal and/or a history of abnormal bleeding or bruising.
* Participant has a history of alcohol or drug abuse within 3 months before screening or excessive alcohol consumption (i.e., > 21 units/week for males, > 14 units/week for females) (1 unit is equal to approximately 1/2 pint [200 milliliters (mL)] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits).

Note: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-08-19 (Actual); Primary Completion 2025-10-25 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Treprostinil (TRE) | Pre-dose and post-dose at multiple timepoints up to Day 10
Area Under Plasma Concentration-Time Curve From 0 to Last Time Point With Quantifiable Concentration (AUClast) of TRE | Pre-dose and post-dose at multiple timepoints up to Day 10
Area Under Plasma Concentration-Time Curve From 0 to Infinity (AUCinf) of TRE | Pre-dose and post-dose at multiple timepoints up to Day 10

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) of TRE | Pre-dose and post-dose at multiple timepoints up to Day 10
Terminal Elimination Half-Life (t1/2) of TRE | Pre-dose and post-dose at multiple timepoints up to Day 10
Apparent Clearance Following Inhalation Administration (CL/F) of TRE | Pre-dose and post-dose at multiple timepoints up to Day 10
Apparent Volume of Distribution at Terminal Phase (Vz/F) of TRE | Pre-dose and post-dose at multiple timepoints up to Day 10
Dose-Normalized Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf/D) of TRE | Pre-dose and post-dose at multiple timepoints up to Day 10
Dose-Normalized Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable (AUClast/D) of TRE | Pre-dose and post-dose at multiple timepoints up to Day 10
Dose-Normalized Cmax and Calculated as Cmax/Dose of TRE | Pre-dose and post-dose at multiple timepoints up to Day 10
Number of Participants Who Experienced at Least One Treatment Emergent Adverse Event (TEAEs) | Up to Day 17

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No